CLINICAL TRIAL: NCT00213967
Title: The Effect of Needle Temperature on Pain Ratings Following Intramuscular Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double
Other Study IDs: 2005-0247
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2008-01

CONDITIONS: Influenza
Keywords: Influenza vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Syringes

INTERVENTIONS:
Device: 22 gauge 1 1/2 inch needles on a 3 ml syringe — cold needles or needles kept at room temperature

SUMMARY:
This study will determine whether decreasing pain associated with intramuscular injection by decreasing needle temperature could be an inexpensive, simple way to decrease injection fear and increase immunization rates.

DETAILED DESCRIPTION:
Influenza virus infection causes significant morbidity and mortality each season. More than 90 million doses of influenza vaccine are administered in most seasons. All of these vaccine doses, except about two million, are administered by intramuscular injection. Surprisingly little research has been done to evaluate appropriate intramuscular injection technique.

A small proportion of the population for which annual influenza immunization is indicated may self-defer because of the pain associated with the administration of the vaccine. Injection is a procedure that causes minor pain. Ice packs are often used for local anesthesia. Decreasing pain associated with intramuscular injection by decreasing needle temperature could be an inexpensive, simple way to decrease injection fear and increase immunization rates.

To test our hypothesis, we will use a double blind controlled study design. Study participants will receive two injections. One injection will contain 0.5ml of next season's influenza vaccine. The other injection will contain 0.5ml normal saline. Each study participant will be randomly assigned to order of injection and to frozen or room temperature needle. (Figure 1) We include two injections to increase the amount of information that we can obtain from the study. In addition to determining if frozen needles decrease discomfort associated with injection of influenza vaccine, we may be able to make our study more generalizable if frozen needles also decrease the pain associated with a normal saline intramuscular injection. Further rationale for the study design covers that we are unable to administer the same injection at two sites to the same person during the same visit varying only the temperature of the needle. To minimize variability, both injections will be administered by the same immunizer who will be blind to the study group assignment. We will maintain blinding of the immunizer by having the person preparing the injections hand the filled syringes to the immunizer uncapped since the immunizer would likely be able to feel the cold of the frozen needles during the needle uncapping. A 1 inch 23 gauge needle (safety injection device; Eclipse by BD, Franklin Lakes, NJ) will be used for all participants under 90kg. A 1 ½ inch needle will be used for all larger participants. We will ask each individual to rate the pain of each injection using a standard 10 point pain scale.1 Each participant will be asked which injection was less painful and if he/she can tell us if a frozen needle was used for either or both injection. Members from the research team will call or email subjects 2-4 days after the administration of the injection. During this phone call, subjects will be asked to rate their current pain at both injection sites. They will also be asked if they notice any redness around the injection site. This additional phone call will help to determine if needle temperature affects delayed injection site reactions (minor soreness and/or redness around the injection site lasting 1-3 days after the injection) in addition to immediate effects.

To determine if there is an effect on influenza vaccine if administered with cold needles, we will measure antibody response to influenza vaccine. Blood will be drawn immediately following the administration of the intramuscular injections and pain scoring from a subset of study participants. Sub-study participants will return in 2-4 weeks for a second blood draw to measure post-immunization antibody concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults

Exclusion Criteria:

* Immunosuppressive medications or medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2005-10; Primary Completion 2006-12 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Pain level

SECONDARY OUTCOMES:
Antibody Response

CONTACTS AND LOCATIONS:
Overall Officials: Mary S Hayney, PharmD, Principal Investigator — University of Wisconsin, Madison